CLINICAL TRIAL: NCT01959789
Title: In-office Bleaching With a 2-day Interval Between Sessions: Tooth Sensitivity
Status: Completed | Type: Observational
Sponsor: Universidade Estadual de Ponta Grossa (Other)
Responsible Party: Principal Investigator, Eloisa Andrade de Paula, Student, Universidade Estadual de Ponta Grossa
Other Study IDs: 22564/2011; name (Registry Identifier: In-office bleaching with a 2-day interval between sessions.); Name of trial (Registry Identifier: In-office bleaching with a 2-day interval between sessions.)
Record Dates: First submitted 2013-10-06; First posted 2013-10-10 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Dentin Sensitivity
Keywords: Randomized Controlled Clinical Trial; Tooth Bleaching
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: Standard treatment
- 2 days: bleaching treatments made in 2 days

SUMMARY:
The calcium containing 35% hydrogen peroxide gel employed in this study can be re-applied 2 days after the first bleaching session without increasing the bleaching-induced tooth sensitivity

DETAILED DESCRIPTION:
The in-office bleaching uses 35% hydrogen peroxide gel which is applied in 2 to 3 sessions usually with one week interval between sessions, without a scientific and plausible reason for this recommendation (. The aim of this study was to evaluate the tooth sensitivity (TS) risk using a shorter interval between clinical sessions. Methods: In this randomized, single-blind study, 40 young patients with color C2 or darker were selected and randomly divided in two groups. In the 7-day group, two bleaching sessions with a 35% hydrogen peroxide gel (Whiteness HP Blue Calcium - FGM) were performed with a one-week interval and in the 2-day group, the same protocol was performed but with a 2-day interval. TS was recorded on a 0-10 visual analog scale up to 48 h after bleaching. The color evaluation was performed at baseline and 30 days after bleaching with a value-oriented shade guide and a spectrophotometer. The absolute risk of TS (%) was evaluated by Fisher´s exact. The TS intensity was evaluated by two-way repeated measured ANOVA and color changes (ΔSGU and ΔE) were evaluated by Student´s t-test (alpha = 5%).

ELIGIBILITY:
Inclusion Criteria:

The participants should have:

At least six maxillary and mandibular anterior teeth caries-free. Without restorations on the labial surfaces. The central incisors should be C2 or darker according to a value-oriented shade guide (Vita Lumin).

-

Exclusion Criteria:

Pre-existing anterior restorations. Pregnant/lactating. Severe internal tooth discoloration (tetracycline stains, fluorosis, pulpless teeth).

Taking any drug with anti-inflammatory and antioxidant action. Bruxism habits or any other pathology that could cause Tooth Sensbility (such as recession, dentine exposure).

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants included in this clinical trial were at least 18 years old and had good general and oral health. Participants were recruited by means of visual communication through posters in the university and in stores at Umuarama city. A total of 116 participants were examined in a dental chair to check if they met the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Tooth sensibility | 1 year

SECONDARY OUTCOMES:
Color | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eloisa A Paula, MD, Principal Investigator — Universidade Estadual de Ponta Grossa
Locations (1):
- Universidade Paranaense - UNIPAR, Umuarama, Paraná, Brazil

REFERENCES:
- [Derived] de Paula EA, Nava JA, Rosso C, Benazzi CM, Fernandes KT, Kossatz S, Loguercio AD, Reis A. In-office bleaching with a two- and seven-day intervals between clinical sessions: A randomized clinical trial on tooth sensitivity. J Dent. 2015 Apr;43(4):424-9. doi: 10.1016/j.jdent.2014.09.009. Epub 2014 Sep 23. PMID 25257824